CLINICAL TRIAL: NCT05919173
Title: UROLOGICAL SURGERIES IN CHILDREN: Comparison Between 0.25% Bupivacaine and 0.25% Bupivacaine withDexmedetomidine in the Caudal Block
Brief Title: Comparison Between Bupivacaine and Bupivacaine With Dexmedetomidine in Caudal Block for Post Operative Pain Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sindh Institute of Urology and Transplantation (Other)
Responsible Party: Principal Investigator, Dr. Shakil Malik, Assistant professor, Sindh Institute of Urology and Transplantation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SIUT-ERC-2021/A-258
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Injections

STUDY DESIGN:
Intervention Model Description: comparative study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupivacaine 0.25% (Experimental): Bupivacaine 0.25% Dose: 1mL/kg body weight
  Interventions: Drug: Bupivacaine Hydrochloride 0.25% Injection Solution
- Bupivacaine+DEX (Experimental): Bupivacaine 0.25% plus Dexmedetomidine 1microgram/kg Dose: 1mL/kg
  Interventions: Drug: Bupivacaine Hydrochloride 0.25% Injection plus Dexmedetomidine 1 microgram/kg body weight

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride 0.25% Injection Solution — Bupivacaine Hydrochloride 0.25% Injection Dose: 1mL/kg (milliliter per kilogram body weight)
  Arms: Bupivacaine 0.25%
Drug: Bupivacaine Hydrochloride 0.25% Injection plus Dexmedetomidine 1 microgram/kg body weight — Bupivacaine HCL 0.25% Injection plus Dexmedetomidine 1micro/kg Dose: 1 mL/kg (milliliter per kilogram body weight)
  Arms: Bupivacaine+DEX

SUMMARY:
The aim of this study is to compare the duration of analgesia, sedation, and intra and postoperative hemodynamics. This drug is recently available in Pakistan. To the best of our knowledge, no published data is available in this respect in Pakistan, so this study would in turn help to fill the gap in knowledge in low-resource settings/emerging economy.

DETAILED DESCRIPTION:
Postoperative pain is an annoying subjective sensation for both children and their parents. Almost 80% of the patients undergoing surgery experience postoperative pain, and 80% of them reported moderate to severe pain intensity. Management of postoperative pain has become a major concern in pediatrics. Results of many studies in different countries show that postoperative pain in children is inadequate. Lee et al showed that one of the main reasons for inadequate treatment of postoperative pain in children is difficulties with pain assessment and concerns related to the side effects of opioid analgesics.

The regional anesthetic technique significantly decreases postoperative pain and systemic analgesic requirements. Caudal block, usually combined with general anesthetic technique is one of the most popular, reliable, and safe anesthesia techniques for abdominal and lower limb surgeries in children but the main disadvantage of caudal analgesia is the short duration of action after a single injection.

Bupivacaine is a long-acting, reliable local anesthetic agent that is used as a caudal analgesic, but different auxiliary agents need to be co-administered to improve its analgesic efficiency. Various additives used in the past to increase the pain-free period postoperatively and to decrease the analgesic requirement such as midazolam neostigmine, ketamine, clonidine, and dexmedetomidine.

Dexmedetomidine is a potent and highly selective alpha 2 adrenergic agonists that has been described as safe and effective in many anesthetic applications and analgesic techniques. In contrast to other agents, it has sympatholytic, analgesic, and sedative effects, and is randomly free from side effects except for manageable hypotension and bradycardia.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 & 2
* elective per-urethral cystolithotripsy

Exclusion Criteria:

* History of developmental delay or mental retardation
* Known or suspected coagulopathy
* Known allergy to any of the study drugs
* Any signs of infection at the site of the proposed caudal block
* Any caudal anatomical deformity

Ages: 2 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Post operative Pain | 24 hour post operatively
  * face, legs, activity, cry, and consolability (FLACC) behavioral pain scale
  * Each category is scored on the 0-2 scale which results in a total score of 0-10.
  * Assessment of FLACC Pain Score:
    * 0 = Relaxed and comfortable
    * 1-3 = Mild discomfort
    * 4-6 = Moderate pain
    * 7-10 = Severe discomfort/pain

CONTACTS AND LOCATIONS:
Overall Officials: Ali A Lanewala, MD, PhD, Study Director — Sindh Institute of Urology & Transplantation
Locations (1):
- Sindh Institute of Urology and Transplantation. Department of Anaesthesia and Surgical Intensive Care Units, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No